CLINICAL TRIAL: NCT06134544
Title: Effect of Isomaltooligosaccharides on Intestinal Bacterial Translocation in Patients With Liver Cirrhosis: a Single-center, Single-arm Study
Brief Title: Effect of IMO on Intestinal Microbiota Translocation in Cirrhosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NFEC-2023-457
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Intervention Model Description: Acutely decompensated cirrhosis ( with ascites).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of IMO (Experimental): Patients will be given IMO (20g/100ml) for 7 days.
  Interventions: Dietary Supplement: Isomaltooligosaccharides (IMO)

INTERVENTIONS:
Dietary Supplement: Isomaltooligosaccharides (IMO) — Patients will still receive standard treatment, including medicine and other invasive treatment.

SUMMARY:
The goal of this intervention clinical trial is to learn about the protection of isomaltooligosaccharides (IMO) on intestinal bacterial translocation in patients with liver cirrhosis. The main question is to answer the changes of LPS after adminstration of IMO.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-75.
* Cirrhotic patients.
* Decompensation event: ascites.
* LPS>0.45EU/ml.

Exclusion Criteria:

* Pregnant or breast-feeding.
* Active bacterial or fungal infection.
* Other decompensations: Hepatic encephalopathy, gastroesophageal varices and hemorrhage.
* Diagnosis of EASL-ACLF.
* Diarrhea.
* Malignancy.
* Anticipated short survival time.
* Adverse reactions or allergies to oral carbohydrate preparations.
* Substance abuse or addiction.
* Severe extrahepatic diseases (e.g. patients with CKD-5 stage, severe cardiopulmonary dysfunction, and psychiatric disorders).
* Be immunosuppressed or immunodeficient states and the use of immunoglobulins or other immune-boosting conditions.
* Be unsuitable for participating in this trial.
* Participated in any drug trial within the past month
* History of antibacterial or fungal use within 1 week prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Lipopolysaccharide (LPS) in plasma | Before (Day-0) and after treatment (Day-8).
  LPS will be tested by Tachypiens Amebocyte Lysate (TAL) test

SECONDARY OUTCOMES:
Changes of bacterial load in plasma | Before (Day-0) ,after treatment (Day-8), after 7-day non-treatment (day 15).
  Count the Colony-Forming Units (CFU) to value the bacterial load
Changes of markers of infections (CRP) in plasma | Before (Day-0) ,after treatment (Day-8), after 7-day non-treatment (day 15).
  C-reactive protein
Changes of markers of infections (PCT) in plasma | Before (Day-0) ,after treatment (Day-8), after 7-day non-treatment (day 15).
  Procalcitonin，PCT
Changes of markers of kidney failure (Cr) in plasma | Before (Day-0) ,after treatment (Day-8), after 7-day non-treatment (day 15).
  Creatinine，Cr
Changes of markers of coagulation failure (INR) in plasma | Before (Day-0) ,after treatment (Day-8), after 7-day non-treatment (day 15).
  International normalized ratio，INR
Changes of markers of liver failure (TBIL) in plasma | Before (Day-0) ,after treatment (Day-8), after 7-day non-treatment (day 15).
  Total bilirubin，TBIL
Changes of Lipopolysaccharide (LPS) in plasma after 7-day non-treatment | After 7-day non-treatment (day 15).
  LPS will be tested by Tachypiens Amebocyte Lysate (TAL) test
Incidence of bacterial infection | After treatment (Day-8) up to follow-up (Day-28)
  All kinds of infection, including pneumonia, SBP, urine tract infection and so on.
Development of acute-on-chronic liver failure | After treatment (Day-8) up to follow-up (Day-28)
  Diagnosis of ACLF is based on the criteria of EASL-ACLF.
Changes of Meld scores which evaluate severity of liver diseases. | Before (Day-0) ,after treatment (Day-8), after 7-day non-treatment (day 15).
  Model for End-Stage Liver Disease (MELD) is used to estimates a patient's chances of surviving their disease during the next three months. This numerical scale is used for adult patients waiting for a transplant. The MELD score ranges from 6 to 40 (gravely ill). The individual score tells you what is the urgency of undergoing a liver transplant during the next 90 days (three months).
28-day mortality | Day-28

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No